CLINICAL TRIAL: NCT03757741
Title: Impact of Inflammation-mediated Myocardial Fibrosis on the Risk of Recurrence After Successful Ablation of Atrial Fibrillation - the FIBRO-RISK Study
Brief Title: Inflammation, Fibrosis and Risk of Recurrence After Atrial Fibrillation Ablation
Acronym: FIBRO-RISK
Status: Completed | Type: Observational
Sponsor: Cardio Med Medical Center (Industry)
Collaborators: University of Targu Mures, Romania (Other); University Hospital of Targu Mures, Romania (Other)
Responsible Party: Sponsor
Other Study IDs: CM0318-FIR
Record Dates: First submitted 2018-11-25; First posted 2018-11-29 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2020-07

CONDITIONS: Atrial Fibrillation; Atrial Inflammation
Keywords: atrial fibrillation recurrence; atrial volume; atrial fibrosis; epicardial adipose tissue; inflammatory biomarkers; late gadolinium-enhancement cardiac magnetic resonance; pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- AF-SG 01: Study subjects with atrial fibrillation recurrence after ablation: Blood sampling (assessment of complete blood count, biochemistry, inflammatory biomarkers), 2D transthoracic echocardiography, Late Gadolinium-Enhancement Cardiac Magnetic Resonance, and complex left and right atrium analysis, Pulmonary vein isolation radiofrequency ablation
  Interventions: Diagnostic Test: Cardiac imaging tests; Diagnostic Test: Venous blood samle collection
- AF-SG 02: Study subjects without atrial fibrillation recurrence after ablation: Blood sampling (assessment of complete blood count, biochemistry, inflammatory biomarkers), 2D transthoracic echocardiography, Late Gadolinium-Enhancement Cardiac Magnetic Resonance, and complex left and right atrium analysis, Pulmonary vein isolation radiofrequency ablation
  Interventions: Diagnostic Test: Cardiac imaging tests; Diagnostic Test: Venous blood samle collection

INTERVENTIONS:
Diagnostic Test: Cardiac imaging tests — 2D transthoracic echocardiography; Late gadolinium-enhancement cardiac magnetic resonance with the evaluation of pulmonary veins anatomy, atrial fibrosis, atrial volumes and the amount of epicardial fat will
Diagnostic Test: Venous blood samle collection — Venous blood sample collection 1 day prior to the ablation procedure: Serum levels of high sensitive C Reactive Protein, Matrix metalloproteases, Interleukin-6, and N-Terminal Pro-B-Type Natriuretic Peptide.

SUMMARY:
FIBRO-RISK study aims to investigate the impact of inflammatory-mediated myocardial fibrosis on the risk of recurrence after successful ablation of atrial fibrillation. The level of systemic inflammation in the pre-ablation and immediate post-ablation period will be assessed on the basis of serum levels of inflammatory biomarkers (hs-CRP, matrix metalloproteases, interleukin-6), while the level of cardiac fibrosis will be determined based on MRI imaging associated with complex post-processing techniques for mapping myocardial fibrosis at the level of left atrium and left ventricle. At the same time, the amount of epicardial fat will serve as an indirect marker of localized inflammation and will be determined at different levels in the heart (surrounding left atrium, right atrium or the entire heart), while ventricular function will be assessed on the basis of serum levels of NT pro-BNP prior to the procedure. All these parameters will be investigated in patients with successful ablation of AF, who will be divided into 2 groups: group 1 - patients who develop AF recurrence at 1-year, and group 2 - patients with no recurrence of AF at 1-year. In all patients, the following biomarkers will be determined: serum levels of inflammatory biomarkers and NT-proBNP at 24 hours and 1 year post-procedure, the amount of myocardial fibrosis at the level of left atrium and left ventricle at baseline +/- 7 days and the amount of epicardial fat surrounding left atrium, right atrium and the entire heart at baseline +/- 7 days.

The primary endpoint of the study will be represented by the rate of AF recurrence at 1-year post ablation, documented by either ECG or Holter monitoring.

The secondary endpoints of the study will be:

* rate of re-hospitalization
* rate of survival without relapse
* rate of major adverse cardiovascular events (MACE rate, including cardiovascular death or stroke)

DETAILED DESCRIPTION:
The prevalence of atrial fibrillation (AF) is on the rise, being the most frequent sustained supraventricular arrhythmia and a health issue by its increased morbidity and mortality. In most of the cases, myocardial tissue located at the level of the pulmonary veins represents the trigger for atrial fibrillation. The pathophysiology of AF is still incompletely understood, several studies suggesting that profibrotic and inflammatory processes have a crucial role in the development of AF. So far the success rate of AF ablation is not very high, reaching 70% in patients with paroxysmal AF and 50% in cases with persistent AF. Several risk factors for the occurrence and recurrence of AF have been described in the literature, including left atrial enlargement, left ventricular dysfunction, epicardial fat volume, and myocardial fibrosis caused by local atrial inflammation. What remains to be investigated is the relationship between these risk factors and the recurrence of AF after radiofrequency catheter ablation using advanced 3D mapping system.

This is a clinical prospective, descriptive, single-center study which will be carried out in the Center of Advanced Research in Multimodal Cardiac Imaging Cardiomed Tirgu Mures, Romania. The duration of the study is 2 years which include the initial screening and the follow-up period for the recurrence of AF.

The study will include 100 subjects suitable for catheter ablation. Imaging biomarkers and laboratory analyses such as high sensitive C Reactive Protein (hsCRP), matrix metalloproteases (MMP), interleukin-6 (IL6) and N-Terminal Pro-B-Type Natriuretic Peptide (NT pro-BNP) will be determined in the first 24 hours after the procedure. The anatomy of pulmonary veins, atrial fibrosis, atrial volumes and the amount of epicardial fat will be evaluated and quantified with late gadolinium-enhancement cardiac magnetic resonance (LGE-CMR). All these parameters will be investigated in patients with successful ablation of AF, who will be divided into 2 groups: group 1 - patients who develop AF recurrence at 1-year, and group 2 - patients with no recurrence of AF at 1-year. In all patients, the following biomarkers will be determined: serum levels of inflammatory biomarkers and NT-proBNP at 24 hours and 1 year post-procedure, the amount of myocardial fibrosis at the level of left atrium and left ventricle at baseline +/- 7 days and the amount of epicardial fat surrounding left atrium, right atrium and the entire heart at baseline +/- 7 days.

The study will be conducted over a period of 2 years, in which patients will be examined at baseline, and will be followed-up for recurrence of AF.

All patients will sign an informed written consent and will be checked for the exclusion criteria prior to enrolment.

Study objectives:

Primary: To investigate the correlation between imaging markers provided by cardiac magnetic resonance (including the degree of left atrial and ventricular fibrosis, left and right atrial volume, epicardial fat tissue volume), inflammatory biomarkers, and the risk of AF recurrence post ablation.

Secondary: To investigate the correlation between structural remodeling of the left and right atrium, epicardial fat tissue volume and serum inflammatory biomarkers in patients with AF.

Study Timeline:

* Baseline (day 0)
* Obtain and document consent from participant on study consent form.
* Verify inclusion/exclusion criteria.
* Obtain demographic information, medical history, medication history, alcohol, and tobacco use history.
* Record results of physical examinations and 12-lead ECG.
* Collect blood specimens (complete blood count, biochemistry and inflammatory biomarkers).
* Imaging procedures: transthoracic 2-D echocardiography, late gadolinium-enhancement cardiac magnetic resonance
* Visit 1 (month 1,3,6,12)
* Record results of physical examinations, 12-lead ECG and medical history.
* Imaging procedures: transthoracic 2-D echocardiography
* Final study visit (month 12)
* Record results of physical examinations, medical history,12-lead ECG and determination of serum levels of inflammatory biomarkers and NT-proBNP
* Imaging procedures: transthoracic 2-D echocardiography
* End-point evaluation.

Study procedures:

* Medical history, clinical examination, laboratory tests (complete blood count, biochemistry, serum level of hs-CRP, MMP, IL6, and NT-pro-BNP);
* 12-lead ECG
* 2D transthoracic echocardiography with measurement of cardiac diameters, volumes, valvular function and regurgitation, pressure gradients, left ventricular systolic and diastolic function and ejection fraction.
* Late Gadolinium-Enhancement Cardiac Magnetic Resonance (LGE-CMR) with the evaluation of left and right atrial volume, the volume of epicardial adipose tissue, the degree of atrial and ventricular fibrosis
* Pulmonary vein isolation radiofrequency ablation with advanced 3D mapping system

Data collection: All the information will be collected in a database that consists of patient's background, medical history, medication, imaging features provided by cardiac ultrasound, Cardiac magnetic resonance and CMR imaging post-processing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-valvular paroxysmal or persistent atrial fibrillation who undergo successful ablation of atrial fibrillation, either by cryoablation or by radiofrequency advanced 3D mapping system;
* Ability to provide informed consent;
* Patients aged at least 18 years;

Exclusion Criteria:

* Patients with valvular atrial fibrillation;
* Patients with acute coronary syndrome in the last 30 days
* Patients in whom atrial fibrillation is presumed to be caused by hyperthyreosis
* Patients with long-standing persistent or permanent atrial fibrillation;
* Unwillingness or incapacity to provide informed consent;
* Allergy to gadolinium contrast media;
* Absolute or relative contraindications to magnetic resonance imaging
* Pregnancy or lactation;
* Women with childbearing potential in absence of any contraceptive treatment
* Renal insufficiency (creatinine greater than 1.5 mg/dL) or renal failure requiring dialysis;
* Active malignancy or malignancy within the last 5 year prior to enrollment;
* Conditions associated with an estimated life expectancy of under 2 years;

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population includes patients from a single center with paroxysmal and persistent atrial fibrillation, meeting inclusion and exclusion criteria and undergoing pulmonary vein isolation radiofrequency catheter ablation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
The rate of AF recurrence after pulmonary vein isolation | 12 months
  The primary outcome measure will be represented by the rate of AF recurrence at 1 year post ablation, documented by either ECG or Holter monitoring.

SECONDARY OUTCOMES:
Rate of re-hospitalization | 12 months
  The secondary endpoints of the study will be: rate of re-hospitalization, rate of survival without relapse, rate of major adverse cardiovascular events (MACE rate, including cardiovascular death or stroke)
Rate of survival without relapse | 12 months
  The secondary endpoints of the study will be: rate of re-hospitalization, rate of survival without relapse, rate of major adverse cardiovascular events (MACE rate, including cardiovascular death or stroke)
Rate of major adverse cardiovascular events (MACE rate, including cardiovascular death or stroke) | 12 months
  The secondary endpoints of the study will be: rate of re-hospitalization, rate of survival without relapse, rate of major adverse cardiovascular events (MACE rate, including cardiovascular death or stroke)

CONTACTS AND LOCATIONS:
Overall Officials: Szilamér Korodi, M.D., Principal Investigator — University of Medicine and Pharmacy of Tirgu Mures, Romania
Locations (1):
- Cardio Med Medical Center, Târgu Mureş, Mureș County, Romania

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available for interested parties.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The IPD sharing frame is starting 6 months after publication.